CLINICAL TRIAL: NCT01870635
Title: Ondansetron Administration to WELL Children With Gastroenteritis Associated Vomiting in Emergency Departments in Pakistan
Brief Title: Ondansetron Administration to WELL Children With Gastroenteritis Associated Vomiting in EDs in Pakistan
Acronym: OWEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Stephen Freedman (Other)
Collaborators: Thrasher Research Fund (Other); Bill and Melinda Gates Foundation (Other); Aga Khan University (Other)
Responsible Party: Sponsor-Investigator, Dr. Stephen Freedman, Associate Professor of Pediatrics; Alberta Children's Hospital Foundation Professor in Child Health and Wellness Alberta Children's Hospital Theme Lead, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSO1026252
Record Dates: First submitted 2013-05-30; First posted 2013-06-06 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Dehydration; Gastroenteritis; Vomiting; Diarrhea
Keywords: Low-middle income country; Dehydration; Intravenous Rehydration; Pakistan
MeSH Terms: conditions — Dehydration; Gastroenteritis; Vomiting; Diarrhea | interventions — Ondansetron; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ondansetron (Experimental): 4 mg oral disintegrating tablet of ondansetron
  Participant weight 8-15 kg = half dose (2mg) Participant weight greater than 15 kg = full dose (4mg)
  Interventions: Drug: Ondansetron
- Placebo (sugar pill) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — Eligible children will receive one weight based (0.13 - 0.26 mg/kg) dose of an oral ondansetron disintegrating tablet. Subsequent therapy will be in accordance with World Health Organization guidelines as dictated by the child's hydration status.
  Other Names: Zofran
  Arms: Ondansetron
Drug: Placebo — Eligible children will receive one dose of an oral disintegrating Placebo (sugar pill) tablet. Subsequent therapy will be in accordance with World Health Organization guidelines as dictated by the child's hydration status.
  Other Names: Sugar Pill
  Arms: Placebo (sugar pill)

SUMMARY:
The primary objective is to determine if the administration of a single dose of oral ondansetron (an anti-vomiting medication), compared to placebo, results in a reduction in intravenous (IV) rehydration therapy in children presenting for emergency department care with vomiting and diarrhea in Pakistan.

DETAILED DESCRIPTION:
Gastroenteritis remains one of the most common causes of morbidity and mortality in children <5 years of age worldwide. A critical factor in the reduction in mortality over the past 30 years has been the introduction of oral rehydration therapy (ORT) for the treatment of dehydration.

However, its use has stagnated in many low- and middle-income countries (LMIC) where many children lack access to alternatives such as intravenous (IV) rehydration. When such children have fluid losses that cannot be replaced orally due to intractable vomiting, death is common. Finding a safe, non-invasive, and effective strategy to reduce vomiting in children would substantially decrease the need for IV rehydration and hence morbidity and mortality in LMICs. Although antiemetic agents are included in the WHO list of Essential Medicines, their use in children with gastroenteritis is not endorsed by the World Health Organization (WHO). Concerns include a lack of evidence that antiemetic agents can improve outcomes and that they are associated with dangerous side effects. However, in high-income settings, studies on ondansetron, an antiemetic agent, have demonstrated that it can reduce vomiting, IV rehydration, and hospitalization. Recent reviews by prominent organizations (e.g. International child Health Review Collaboration; the Committee on the Selection and Use of Essential Medicines) have indicated an interest in ondansetron use in children with gastroenteritis, and they have concluded that further evidence is required. This trial aims to determine if the administration of a single dose of oral ondansetron results in improved outcomes in children brought for emergency department care with vomiting and diarrhea in Pakistan.

Two trials will be conducted under the umbrella of one study. The proposed trials will be identical with the exception of the severity of dehydration at enrollment (either "some" or none "well"). The trials will have the following specific aims:

1. To determine, in children 6 - 59 months of age with AGE with vomiting and diarrhea who have "NO" dehydration, if there is a reduction in the proportion of children administered IV rehydration in those who receive oral ondansetron in addition to all WHO standards of care, compared to those receiving an oral placebo in addition to all WHO standards of care.
2. To determine, in children 6 - 59 months of age with AGE with vomiting and diarrhea who have "SOME" dehydration, if there is a reduction in the proportion of children administered IV rehydration in those who receive oral ondansetron in addition to all WHO standards of care, compared to those receiving an oral placebo in addition to all WHO standards of care.

IV rehydration is a powerful marker of treatment failure and reducing the need for IV rehydration therapy in either of these 2 groups of children will be viewed as a significant advance by healthcare providers and decision makers. Previous studies of ondansetron have not been conducted in low and middle income countries (LMIC), have been of relatively small sample sizes, have not employed WHO dehydration scales, and have not focused on young children (i.e. <5 years). As such therapy is unavailable to a large number of children in LMIC countries, the ability to demonstrate that ondansetron can reduce the use of IV rehydration will provide compelling evidence that this drug has the potential to save lives around the world. We postulate that oral ondansetron administration to children in LMIC, if beneficial in our study population, could serve as a feasible and reliable intervention that is available for provision by non-hospital based, outreach, and healthcare providers in remote regions of the world.

This study may have immediate impact on patient management. Based on the results, it will be discovered if oral ondansetron plays a role in reducing the need for intravenous rehydration in children with gastroenteritis in Pakistan. As ondansetron is now available in generic formulations, and is relatively inexpensive, it is anticipated that if this study is positive, ondansetron will be considered for inclusion in the WHO - gastroenteritis care package. This could ultimately lead to a decrease in the need for intravenous rehydration in children in countries such as Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 - 59 months (0.5 - 5 years)
* Symptoms consistent with gastroenteritis (must have a & b)

  1. 1 episode of nonbilious, nonbloody vomiting within the 4 hours preceding triage The requirement for only 1 vomiting episode is based on prior work which similarly required 1 vomiting episode within 4 hours of triage. The later study reported a 17% absolute reduction in the use of IV rehydration. The vast majority of children seeking care and enrolled in the aforementioned study had a significantly greater number of vomiting episodes in the preceding 24 hour (mean >9 episodes).
  2. Presence of ≥ 1 episode of diarrhea during the illness We require the presence of only 1 diarrheal stool to enhance our probability of enrolling children with enteritis (as opposed to other diagnoses). In fact, of the 8 RCTs performed using antiemetics in children with gastroenteritis in developed countries, only 1 even required the presence of any diarrhea as part of the eligibility criteria (and that study required a single diarrheal stool).
* Presence of NO dehydration (NO=not enough signs to classify as some or severe dehydration)

Exclusion Criteria:

* Weight <8 kg
* Vomiting or diarrhea for > 7 days
* Malnutrition: The World Health Organization (WHO) definition will be employed - weight for height below -3z scores of the median WHO growth standards
* Severe dehydration (WHO criteria) or hypotension defined as a systolic blood pressure <70 mm Hg in infants 1 month to 12 months, < 70 mm Hg + (2 x age in years) in children 1-10 years, < 90 mm Hg in children ≥ 10 years
* Prior abdominal surgery (excluding hernia)
* Bilious or bloody vomitus
* Known hypersensitivity to ondansetron or any serotonin receptor antagonist
* History or family history of prolonged QT syndrome
* Taking apomorphine or any medication that is generally accepted as having a risk of causing torsades de pointes
* Patients previously enrolled in the study
* Follow-up will not be possible

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 625 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Intravenous (IV) Rehydration | within 72 hours of randomization
  IV rehydration is defined as the IV administration of ≥20 ml/kg over 4 hours of an isotonic fluid for the purpose of rehydration within 72 hours of randomization. This definition allows for the occurrence of the primary outcome in children who receive maintenance plus replacement of losses and not simply those who receive a fluid bolus. This will not include those who simply receive maintenance fluids (e.g. 4 ml/kg/hr for those weighing < 10 kg). This will also enable us to exclude children who undergo IV insertion for the purpose of medication administration. IV rehydration is a powerful marker of treatment failure, a decrease in which is likely to impact practice and influence decision makers since it is drastically more expensive that ORT, it is painful and is associated with a greater risk of adverse events.

SECONDARY OUTCOMES:
The proportion of children who vomit during the 4 hour observation period | within 4 hour observation period after randomization
The frequency of vomiting during the 4 hour observation period | within 4 hour observation period after randomization
Hospitalization > 24 hours | 72 hours after randomization; 24 hour follow up as needed; chart review 21 days after enrollment
  Total length of stay from Emergency Department (ED) arrival until discharge of > 24 hours, regardless of whether time is spent in the ED or inpatient unit
Volume of Oral Rehydration Solution (ORS) consumed (ml/kg) during the 4 hour observation period | within 4 hour observation period after randomization
Development of "SOME" dehydration during the 72 hours following randomization amongst children who are discharged | within 72 hours of randomization
  All children will be presumed to not be dehydrated at the time of discharge regardless of severity of dehydration at the time of ED presentation.
  SOME Dehydration = 2 or more of the following signs:
  * Restlessness, irritability
  * Sunken Eyes
  * Drinks eagerly, thirsty
  * Skin pinch goes back slowly
Number of diarrheal stools during the 72 hours following randomization | within 72 hours of randomization
  Diarrheal stools are defined, in keeping with the WHO definition as "loose or liquid stools"
Treatment failure | 72 hours after randomization; 24 hour follow up as needed; chart review 21 days after enrollment
  This aggregate outcome will include children who experience the following:
  1. IV rehydration as defined in primary outcome
  2. Nasogastric rehydration for > 24 hours - this implies a failure of outpatient Oral Rehydration Therapy (ORT)
  3. Death within 72 hours (from any cause; in or out of hospital)
Response based on infectious etiology (i.e. bacterial vs. viral), duration of illness (i.e. < 48 vs. ≥ 48 hours), and age (< 18 months vs. ≥ 18 months) | 72 hours after randomization; 24 hour follow up as needed; chart review 21 days after enrollment

OTHER OUTCOMES:
Major Side Effects | 72 hours after randomization; 24 hour follow up as needed; chart review 21 days after enrollment
  Uncommon events such as: Arrythmia and Death. This data is critical to estimate a safety profile of ondansetron in low to middle income countries
Semi- and Intensive Care Unit Admission | 72 hours after randomization; 24 hour follow up as needed; chart review 21 days after enrollment
  This data is critical to estimate a safety profile of ondansetron in low to middle income countries

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MD, Principal Investigator — University of Calgary; Zulfiqar Bhutta, MD, Principal Investigator — Aga Khan University - World Health Organization; Sajid B Soofi, MD, Principal Investigator — Aga Khan University
Locations (2):
- Pakistan (2):
  - Aga Khan University Hospital, Karachi
  - Aga Khan Hospital for Women and Children (AKHWC), Kharadar, Karachi

REFERENCES:
- [Derived] Freedman SB, Soofi SB, Willan AR, Williamson-Urquhart S, Ali N, Xie J, Dawoud F, Bhutta ZA. Oral Ondansetron Administration to Nondehydrated Children With Diarrhea and Associated Vomiting in Emergency Departments in Pakistan: A Randomized Controlled Trial. Ann Emerg Med. 2019 Mar;73(3):255-265. doi: 10.1016/j.annemergmed.2018.09.011. Epub 2018 Nov 2. PMID 30392735